CLINICAL TRIAL: NCT02138656
Title: The Effectiveness of Chiropractic in the Treatment of Infantile Colic
Brief Title: CHiropractic for Infantile Colic Study
Acronym: CHIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Review of recruitment methods
Sponsor: University of Southampton (Other)
Collaborators: McTimoney College of Chiropractic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ERGO 4866
Record Dates: First submitted 2014-04-28; First posted 2014-05-14 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Infantile Colic
Keywords: Crying; Chiropractic; Infant; pediatric; Infantile colic; Clinical Trial
MeSH Terms: conditions — Colic; Crying | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Best standard care only - not blind (Active Comparator): Best Standard Care (as defined by Map of Medicine care pathway) - counseling and advice.
  Parents aware that infant is not receiving chiropractic treatment
  Interventions: Other: Best Standard Care
- Best Standard Care and Sham - Blind (Sham Comparator): Best Standard Care (as defined by Map of Medicine care pathway) - counseling and advice plus sham chiropractic treatment. Parents unaware of whether infant is receiving real treatment or sham.
  Interventions: Other: Best Standard Care
- BSC & Chiropractic - Not blind (Experimental): Best Standard Care (as defined by Map of Medicine care pathway) - counseling and advice plus real chiropractic treatment.
  Parents aware that infant is receiving chiropractic treatment.
  Interventions: Other: Chiropractic; Other: Best Standard Care
- BSC & Chiropractic - Blind (Experimental): Best Standard Care (as defined by Map of Medicine care pathway) - counseling and advice plus real chiropractic treatment.
  Parents not aware that infant is receiving chiropractic treatment.
  Interventions: Other: Chiropractic; Other: Best Standard Care

INTERVENTIONS:
Other: Chiropractic — Chiropractic treatment delivered in accordance with clinical protocols developed and agreed with the participant clinicians
  Arms: BSC & Chiropractic - Blind; BSC & Chiropractic - Not blind
Other: Best Standard Care — Counselling and advice delivered in accordance with the Map of Medicine care pathway for Infantile colic

SUMMARY:
The purpose of this study is to investigate whether a course of chiropractic treatment has a significant impact on the natural course of infantile colic, specifically:

1. Do parents of colicky infants randomised to the groups receiving a course of McTimoney chiropractic treatment:

   * report a significantly greater improvement in hours of crying than those in the control group?
   * report a significantly greater improvement their own quality of life (anxiety and depression)?
   * report "resolution" of colic following treatment than the control group?
2. What effect does parental blinding have on parentally-reported symptoms of infantile colic and parental quality of life?

The study will also include exploratory investigations to determine whether there are:

1. Any particular groupings of patient characteristics (for example; 'other' presenting symptoms, position in the natural course of colic, age of onset, spinal dysfunction, perinatal factors) that are associated with good or poor outcomes
2. Any particular characteristics of the treatment (e.g. specific adjustments) that are associated with good or poor outcomes.

DETAILED DESCRIPTION:
Overall Design

The study will be a two-by-two factorial design combining groups of chiropractic treatment or 'Best Standard Care' with blinded or unblinded parents.

The two treatment groups will be 'Best Standard Care only' (BSC) and 'Best Standard Care plus chiropractic' (Chiro). Best standard care will be based on the recommendations from United Kingdom (UK) National Health Service (NHS), using the Map of Medicine care map. Chiropractic treatment will be delivered according to the protocol defined by the participating chiropractors.

There will be two blinded and two unblinded groups. The blinded BSC group will receive the 'sham' treatment in addition to the BSC counselling. The unblinded BSC group will not require this.

In addition, to allow the effects of the n-shaped curve inherent in the natural course of colic to be evaluated, all groups will be stratified by age at entry (below 4 weeks (expected increasing crying over the 2 weeks of the main intervention), between 4 and 6 weeks (expected plateau), and over 6 weeks (decreasing crying)).

The study has a longitudinal design over a ~4 1/2 week period.

For the primary outcomes which take data from the crying diaries, the main data points are defined as:

* Baseline: the 24 hour period of the day before the first treatment
* First treatment: the 24 hour period of the day after the first treatment
* Mid-point treatment: the 24 hour period of the day after the second treatment
* Final treatment: the 24 hour period of the day after the third treatment

Secondary outcomes will include data from the following points:

* Follow-up 1: the 24 hour period of the day 7 days after the third treatment
* Follow-up 2: the 24 hour period of the day 14 days after the third treatment

Other data will be sourced from:

* The initial visit questionnaires
* Follow-up questionnaires approximately 2 days after first treatment, 2 days after 2nd treatment, 2 days after final treatment, around day 21 and day 28.

Instruments

Data collection will be done through 8 main data collection instruments, drafts of which have now been developed:

* First contact questionnaire
* Crying Diary (including severity of other symptoms)
* Initial Visit Questionnaire - Part 1 (demographics and history)
* Initial Visit Questionnaire - Part 2 (success of blinding)
* Credibility and Expectancy Questionnaire (CEQ)
* Hospital Anxiety and Depression Scale
* Adjustments record
* Weekly telephone questionnaire

Power

The sample size is 160, calculated achieve 80% power, 5% significance level, and using an estimated standard deviation of around 2 (based on results from similar studies) for a 1 hour between-groups difference (identified as a 'clinically relevant reduction in crying time' from a parental survey) and allowing for a 25% attrition rate in the latter 2 weeks (based on experiences in similar studies).

Analysis:

Primary Outcomes

For the primary analyses comparisons will be carried out using all the data in one analysis which will assess the significance of the treatments, the blindness and the age groups in an ANCOVA. This will include interaction terms to assess whether the treatment effects are different for the different levels of blindness and for the different age groups and all baseline variables will be included as covariates.

A logistic regression analysis will be used to produce odds ratios for the comparison of treatment, blindness and age groups. The between-groups differences in proportion (risk ratio) of patients reporting 'complete resolution' of colic symptoms (PGIS) after first, mid-point and final treatments (primary outcome) and at follow ups (secondary outcomes) Adverse events will be reported with no analysis. Extraction of primary data from crying diaries will be performed by observers blinded to group allocation.

The primary analysis will be performed by a statistician blinded to group allocation.

Secondary Outcomes

The primary analysis of primary outcomes will be extended to days 21 and 28, as above.

The ANCOVA will be extended to evaluate the between-group differences in

* Cost of NHS resource usage
* Duration that the infant is fussy It is anticipated that parent compliance in completing the diary is likely to deteriorate during once the clinic visits have ceased. However, regular telephone calls will attempt to encourage continued completion. The primary study outcomes will be based on the first 15 days of the diary and it is anticipated that there will be greater compliance during this time.

Investigative Analysis

The exploratory investigations seek to establish any associations between the outcome measures (daily hours crying, presence of other symptoms, Parental Global Impressions of Severity (PGIS), Parental Global Impressions of Change (PGIC), and 'resolution' of colic) after first, mid-point and final treatments, and at follow-ups and any other predictor variables as gathered in the initial visit (Part 1). For example, :

* baseline daily hours crying
* initial symptom trajectory; worsening, plateau, improving
* baseline 'other symptoms' not at all, low, medium and high severity
* age at onset
* perinatal factors (Miller, 2007)
* treatment characteristics

Intention to treat v per protocol

Since this is a clinical study, the primary analysis will be done on an intention-to-treat basis, including any patients who fail to comply with the protocol for their group (e.g. dropping out of the treatment groups).

For some of the analyses, accurate data is required (e.g. actual adjustments performed) which cannot be imputed. In these cases, the analysis will be done on a per protocol basis.

Missing data

Previous studies have reported that the majority of dropouts occur in the no-treatment groups due to worsening symptoms and in the treatment groups due to resolution of symptoms, so data imputed at last value carried forward will represent a conservative approach. For the primary crying time outcome data, where there is a record for Day 8, this will be carried forward to Day 15.

Where reasons for withdrawal on the basis of worsening symptoms are given, this will be included as data points within the PGIS & PGIC analysis, so no imputation will be required.

Attempts will be made to contact any drop-outs to ascertain their reasons for choosing not to continue in the study and these will be reported separately.

For the other analyses, a longitudinal analysis of variance will assess changes over time for the treatment, blindness and age groups together with any interactions and covariates. Although there may be some loss of data in the later time periods, a repeated measures analysis should be able to cope with this without imputation of missing data.

Numbers of subjects responding to the study and progressing to each stage will be recorded on a CONSORT-style flow diagram.

ELIGIBILITY:
Inclusion Criteria:

* Parentally-reported crying of more than three hours per day for three or more days in the preceding week (reported at initial contact to determine preliminary diagnosis of colic)
* Confirmation at first clinic visit that the infant has cried for more than three hours per day for at least one day in the base-lining period.
* Otherwise normal infants, born at term, with normal growth and development, and no indication of other underlying pathology
* Parents fluent in English, providing informed written consent

Exclusion Criteria:

* Infants who have received previous chiropractic, osteopathic or other manipulative treatment

Ages: 1 Day to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes to the duration of crying per day | Baseline to day after first clinic visit (~day 2), mid point (~day 8) and final clinic visit (~day 15)
Proportion of infants achieving clinically-relevant reduction in crying time | Baseline to day after first clinic visit (~day 2), mid point (~day 8) and final clinic visit (~day 15)
  Defined as 60 minutes (median) based on survey
Proportion of infants reported with absence of 'colic' | Follow-up telephone call after first, mid point and final clinic visit (approx days 2, 8 and 15)
  Taken from the Parental Global Impression of Severity scale
Number of adverse events | at any time during an infant's engagement in the study, circa 28 days

SECONDARY OUTCOMES:
Changes to the duration of crying per day | baseline to day 21 and day 28
Changes to parental anxiety and depression scores | first visit (day 1) to each of the 5 follow-up questionnaires (~day 2, 8, 15, 21 & 28)
Proportion of infants achieving clinically-relevant reduction in crying time | From baseline to day 21 and day 28 follow ups
Proportion of infants reported with absence of 'colic' | At day 21 and day 28 (final 2 follow-ups)
Parental Global Impressions of Change in symptoms | At each of the follow-up questionanaires (~day 2, 8, 15, 21 and 28)
Cost of NHS resources used | Reported 'during the preceding week' at each telephone questionnaire (~day 2, 8, 15, 21 and 28)
  Costs calculated based on reported interactions and standard costs published annually by the Personal Social Services Research Unit (PSSRU) in the UK.
Change to Severity of colic-related specific symptoms | Baseline to day after first, mid point and final clinic visits (~days 2, 8, 15) then to day 21 and day 28
  Based on 5-point likert scale 'not at all' to 'a very great deal' for crying with high pitched sound, crying with pain cry, pulling faces (apparently in pain), having a flushed face, holding breath, clenching fists, bending elbows/holding arms rigid, punching fists, wind milling arms, kicking legs, drawing legs up, arching back, tense/distended abdomen, borborygmus, flatulence, vomiting/regurgitating
Change to Parental Global Impressions of Severity | Baseline to follow-ups after first second and final clinic visits (~days 2, 8, 15) then to day 21 and day 28 follow ups
Effectiveness of Blinding | immediately after first "treatment" (day 1) and at follow-up telephone questionnaires after first, mid point and final clinic visits (~day 2, 8 and 15)
  Proportion of correct, incorrect and 'don't know' guesses, reported using James' and Bangs' blinding indices

CONTACTS AND LOCATIONS:
Overall Officials: George Lewith, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom